CLINICAL TRIAL: NCT04112264
Title: Effect of Monopolar Radiofrequency Ablation for Genicular Nerves Compared to Bipolar Radiofrequency Ablation Using Ultrasound in Treating Chronic Knee Osteoarthritis
Brief Title: Ultrasound-guided Monopolar Versus Bipolar Radiofrequency Ablation for Genicular Nerves in Chronic Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD.19.03.152
Record Dates: First submitted 2019-09-25; First posted 2019-10-02 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Chronic Knee Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monopolar radiofrequency ablation (Experimental): Patients will receive ultrasound-guided monopolar radiofrequency ablation
  Interventions: Procedure: Monopolar radiofrequency ablation
- Bipolar radiofrequency ablation (Active Comparator): Patients will receive ultrasound-guided bipolar radiofrequency ablation
  Interventions: Procedure: Bipolar radiofrequency ablation

INTERVENTIONS:
Procedure: Monopolar radiofrequency ablation — a radiofrequency cannula is advanced under USG guidance towards the nerve. The final position will be confirmed by using nerve stimulator with elicitation of paraesthesia along the area of knee joint supplied by that respected genicular nerve by stimulation at 50 Hz current of <0.5 mV. The motor stimulation will be negative at all instances. For each genicular nerve, two conventional RF lesions are done for 120s at 80° of temperature using the Neurotherm 1100 RF generator.
  Arms: Monopolar radiofrequency ablation
Procedure: Bipolar radiofrequency ablation — Two radiofrequency cannula are advanced under USG guidance towards the nerve. The final position will be confirmed by using nerve stimulator with elicitation of paraesthesia by stimulation at 50 Hz current of <0.5 mV. The motor stimulation will be negative at all instances. For each genicular nerve, two conventional RF lesions are done for 120s at 80° of temperature using the Neurotherm 1100 RF generator.
  Arms: Bipolar radiofrequency ablation

SUMMARY:
Radiofrequency ablation of the genicular nerves using ultrasound is safe and effective for treating intractable knee osteoarthritis pain by using either monopolar or bipolar radiofrequency ablation.

This technique is based on anatomical studies demonstrating that genicular nerves are accompanied by genicular arteries. Ultrasound-guided RF genicular ablation yielded both significant reductions in knee pain and improvements in functional capacity.

DETAILED DESCRIPTION:
The aim of this study is to compare between ultrasound guided monopolar and bipolar radiofrequency ablation in chronic knee osteoarthritis.

Osteoarthritis of knee joint is one of the most common disease conditions with advanced age and leads to considerable morbidity in terms of pain, stiffness, limitation in functions, disturbance in sleep and psychological disturbance

A diagnostic genicular nerve block (GNB) with local anesthetic is performed before RF genicular ablation, and a successful response to GNB is considered to indicate the need for RF genicular ablation

ELIGIBILITY:
Inclusion Criteria:

* Radiologic tibiofemoral Osteoarthritis (Kellgren-Lawrence grade 2-4).
* Patients not responding to other treatments as physiotherapy, oral analgesics, and intraarticular injection with hyaluronic acids or steroids.
* Patients refused surgery.

Exclusion Criteria:

* Patient refusal.
* Prior knee surgery.
* Acute knee pain.
* Intra-articular knee corticosteroid or hyaluronic acid injection in the past 3 months.
* Connective tissue diseases that affected the knee.
* Anticoagulant medication use.
* Local skin infection and sepsis at the site of intervention

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-04 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Osteoarthritis pain | basal value, at 1, 4, 12, 24 weeks post procedure
  The mean changes from baseline levels of osteoarthritis pain using visual analogue scale used to measure pain intensity. It is 10 cm scale where 0 cm represent no pain and 10 cm represent the worst pain ever

SECONDARY OUTCOMES:
Oxford Knee Score | basal value, at 1, 4, 12, 24 weeks post procedure
  A specific score to assess the functional changes in the knee using Oxford Knee Score (OKS). The scores are 12-item questionnaires ranging from 12-60, with 12 representing the optimal outcome.
The procedure time | from the start of advancement of the cannula to end of procedure.
  The procedure time taken by each mode of radiofrequency from the start of advancement of the cannula under US guidance to the end of the procedure.
Patient satisfaction score | up to 24 weeks post procedure
  Patient satisfaction score with treatment which is scored from 1 to 10. A score of 1-4 was considered "dissatisfied," 5-8 was "satisfied," and 9 or 10 was "very satisfied
Changes in doses of rescue analgesics | up to 24 weeks post procedure
The incidence of numbness | up to 24 weeks post procedure
The incidence of paresthesia | up to 24 weeks post procedure
The incidence of motor weakness | up to 24 weeks post procedure
the proportion of successful responders | up to 24 weeks post procedure
  the proportion of successful responders with a reduction of at least 50% of median VAS score and no increase from baseline OKS

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Mousa, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol Statistical analysis plan Informed consent form
Time Frame: data will be available at the end of study
Access Criteria: data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement